CLINICAL TRIAL: NCT02756156
Title: Low Dose Interscalene and Infraclavicular Block for Humerus Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Bora Bilal, Assist prof, Kahramanmaras Sutcu Imam University
Other Study IDs: 76263
Record Dates: First submitted 2016-03-15; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-03

CONDITIONS: Humerus Fracture
Keywords: interscalene; infraclavicular; humerus surgery
MeSH Terms: conditions — Humeral Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Combining interscalene block with infraclavicular block for humerus surgery provides a unique surgical anaesthesia and postoperative analgesia.

DETAILED DESCRIPTION:
Interscalene block provides effective surgical anaesthesia for shoulder and proximal arm surgery. However, sometimes it can be inadequate for distal arm surgery. Combining infraclavicular block with interscalene block may provide a successful surgical anaesthesia for humerus surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepting peripheral nerve block technique for humerus surgery
* Unilateral orthopedic humerus surgery
* 18 years of age or older

Exclusion Criteria:

* Patients refused peripheral nerve block
* Non-cooperate patients
* Neuropathy of any etiology in the affected extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing humerus surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Success rate of block | 10 min.- 20 min.
  A complete sensory loss in distribution of the radial, median, ulnar, musculocutaneous and medial cutaneous nerves of the arm

SECONDARY OUTCOMES:
Technique duration | 5 min.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 hours
Complication rate | 24 hours

IPD SHARING:
Plan to Share IPD: No